CLINICAL TRIAL: NCT04295915
Title: Clinical Performance and Reproducibility of the Accelerate PhenoTest™ BC Kit Using the Accelerate Pheno™ System With New Antibiotic Wave I Updates for Antimicrobial Susceptibility Testing of Positive Blood Culture Specimens
Brief Title: Clinical Performance and Reproducibility of the Accelerate PhenoTest™ Blood Culture (BC) Kit With New Antibiotic Wave I Updates
Status: Completed | Type: Observational
Sponsor: Accelerate Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP000026
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Bacteremia
Keywords: Positive blood culture
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Specimens that meet inclusion criteria
  Interventions: Device: Specimens that meet inclusion criteria

INTERVENTIONS:
Device: Specimens that meet inclusion criteria — Specimens that have been de-identified and considered remnant by the laboratory (fresh specimens) or were contrived by the laboratory (using bacterial isolates with no identifying information) can be enrolled into the study.

SUMMARY:
This is a performance and reproducibility study to validate new or updated antimicrobials on the Accelerate PhenoTest™ BC kit. The data from this study will be used to support the submission to the FDA for clearance in the US and for global registrations of the device intended for in vitro diagnostic use.

DETAILED DESCRIPTION:
This clinical study entitled "Clinical Performance and Reproducibility of the Accelerate PhenoTest™ BC Kit Using the Accelerate Pheno™ System with New Antibiotic Wave I Updates for Antimicrobial Susceptibility Testing of Positive Blood Culture Specimens" is designed to demonstrate the clinical performance and reproducibility of the new or updated antimicrobials on the Accelerate PhenoTest™ BC kit, which was previously FDA-cleared in February 2017.

Clinical performance and reproducibility evaluations will be conducted at a minimum of three sites to determine the clinical performance of the new or updated antimicrobials from a combination of fresh (de-identified, remnant specimens) and contrived positive blood culture samples, to include at least 375 total specimens.

The study sites selected will have expertise in blood culture diagnostics and will be able to conduct the study in accordance with this protocol and Good Clinical Practices (GCP). Additionally, prior to study initiation, each site will have approval from the local Institutional Review Board (IRB).

It is anticipated that the data from this study will be used to support the submission to the FDA for clearance in the US and for global registrations of the device intended for in vitro diagnostic use.

ELIGIBILITY:
Inclusion Criteria:

* Blood culture positivity is ≤ 8 hours prior to initiation of testing with the Accelerate Pheno™ system
* Positive blood culture sample containing gram-negative rods according to Gram stain results
* For fresh specimens, de-identified, remnant positive blood culture specimens from patients for which Standard of Care (SOC) testing has been initiated and the remaining samples would otherwise be discarded
* A minimum sample volume of 2.0 mL
* Seeded blood culture specimens derived from archived bacterial

Exclusion Criteria:

* Blood culture positivity is > 8 hours prior to initiation of testing with the Accelerate Pheno™ system
* Insufficient (less than 2.0 mL) remnant sample volume
* From a patient that has already been enrolled in the study
* Fresh samples from Mycobacterial-type blood culture media (BACTEC™ Myco/F Lytic, BacT/ALERT® MP Bottle, VersaTREK® Myco) or charcoal-containing media
* Seeded specimens that appear mixed (by Gram stain or purity plating) after bottle culture positivity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinical or contrived (seeded bacterial isolate) specimens that are indicated as positive by blood culture monitoring systems utilized by clinical microbiology laboratories.
Sampling Method: Non-Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Essential and categorical agreement with Clinical and Laboratory Standards Institute (CLSI) broth microdilution reference method | Approximately 4 months

SECONDARY OUTCOMES:
Essential agreement of MICs compared to the modal MIC values obtained for intra- and inter-laboratory results | Approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Campeau, Study Director — Accelerate Diagnostics, Inc.
Locations (3):
- United States (3):
  - Accelerate Diagnostics, Tucson, Arizona
  - Penn State-Hershey Medical Center, Hershey, Pennsylvania
  - Quest/med fusion, Lewisville, Texas

IPD SHARING:
Plan to Share IPD: No